CLINICAL TRIAL: NCT05684614
Title: Interoception and Emotion Regulation in Healthy Individuals
Brief Title: Interoception and Emotion Regulation
Acronym: INTEROEMOTION3
Status: Completed | Type: Observational
Sponsor: University of Valencia (Other)
Responsible Party: Principal Investigator, Rosa M. Baños Rivera, Full Professor, University of Valencia
Other Study IDs: 1533450; FPU18/01690 (Other Grant/Funding Number: Ministerio de Ciencia e Innovación)
Record Dates: First submitted 2022-12-06; First posted 2023-01-13 (Actual); Last update posted 2023-12-12 (Actual); Status verified 2023-12

CONDITIONS: Mood Change; Emotion Regulation
MeSH Terms: conditions — Emotional Regulation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Healthy individuals: Adult individuals recruited from the community through announcements at the university and social media
  Interventions: Other: Negative mood induction procedure; Other: Spontaneous emotion regulation task; Other: Positive mood induction procedure

INTERVENTIONS:
Other: Negative mood induction procedure — The negative mood induction procedure (MIP) used in this study has previously been shown to effectively induce sadness. This MIP takes place in a virtual environment of an urban park and includes the following methods to induce negative mood: 1) Velten's tasks, consisting of interactive phrase formulations with negative thoughts and beliefs about the self (e.g., "I don't have any future"); 2) visualizing International Affective Pictures; and 3) recalling a negative autobiographical memory related to a significant loss (e.g., a person, a pet).
Other: Spontaneous emotion regulation task — Participants are instructed to use whatever strategy they want by doing, saying, and/or thinking whatever they want to feel better for 2 min
Other: Positive mood induction procedure — The positive mood induction procedure (MIP) used in this study has previously been shown to effectively induce sadness. This MIP takes place in a virtual environment of an urban park and includes the following methods to induce positive mood: 1) Velten's tasks, consisting of interactive phrase formulations with positive thoughts and beliefs (e.g., "Life is wonderful"); 2) visualizing International Affective Pictures; and 3) recalling a positive autobiographical memory

SUMMARY:
The goal of this observational study is to examine the role of interoception in emotion regulation of negative mood in healthy individuals.

Participants will fulfill several questionnaires and perform the Heartbeat Counting Task. Then, they will receive a negative mood induction procedure, after which they will be instructed to perform a spontaneous emotion regulation task. The mood will be assessed before and after the induction, as well as after the emotion regulation task. It is expected that greater interoceptive abilities will show a greater reduction of negative mood after the emotion regulation task than individuals with lower interoceptive abilities.

DETAILED DESCRIPTION:
This study aims to examine the role of interoceptive abilities in the use of emotion regulation strategies and the success of emotion regulation in regulating the negative mood in healthy individuals. First, it is expected that better interoceptive functioning (namely, higher interoceptive accuracy and interoceptive sensibility) will facilitate the use of adaptive emotion regulation strategies (vs. maladaptive emotion regulation strategies) to regulate the negative mood. In addition, it is expected that individuals with greater interoceptive abilities will show greater efficacy in the emotion regulation process (i.e., greater reduction of negative mood after the emotion regulation task) than individuals with lower interoceptive abilities. However, it is hypothesized that interoceptive abilities will not be related to the induced negative affect.

The whole study is conducted in one single 1-hour session. First, participants will be screened to check eligibility inclusion/exclusion criteria. Second, eligible participants will complete baseline measures, namely, trait emotion regulation abilities and interoceptive abilities. Third, participants will complete a mood rating scale, after which they will be applied a negative mood induction procedure (MIP) that has previously been shown to effectively induce sadness. During this MIP, the heart rate variability will be recorded. Next, participants will complete the mood rating scale again. Later, they will perform a spontaneous emotion regulation task. In this task, participants will have 2 min to do, say, and/or think about whatever they need to feel better. Afterwards, participants will again rate their mood and complete the final measures regarding state emotion regulation. Finally, participants will receive a positive MIP (while recording their heart rate variability) and be debriefed. The study will be conducted following the principles stated in the Declaration of Helsinki.

ELIGIBILITY:
Inclusion Criteria:

* Aged above 18
* Absent symptoms of depression as described by scores ≤ 8 in the depression dimension of the Hospital Anxiety and Depression Scale (HADS) (Terol-Cantero et al., 2015; Zigmond & Snaith, 1983)
* Not having cognitive, psychiatric, or neurological impairments (self-reported by participants)

Exclusion Criteria:

* History of/current substance abuse
* A medical condition that prevents participation in this study
* History of traumatic event exposure as self-reported.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The sample in this study will represent a population of neurotypical individuals.
Sampling Method: Non-Probability Sample
Enrollment: 117 (Actual)
Dates: Start 2022-09-06 (Actual); Primary Completion 2023-03-13 (Actual); Study Completion 2023-03-13 (Actual)

PRIMARY OUTCOMES:
Change in Mood before the negative induction, after the negative induction, and after the emotion regulation task | The whole study is conducted in a single experimental session: immediately before the negative mood induction procedure, immediately after the negative mood induction procedure, immediately after the emotion regulation task
  Sadness and joy dimensions of the Scale for Mood Assessment, with scores ranging from 0 to 10, where higher scores indicate higher levels of joy and sadness, respectively.

SECONDARY OUTCOMES:
State difficulties in emotion regulation after the emotion regulation task | The whole study is conducted in a single experimental session: Immediately after the emotion regulation task
  State Difficulties in Emotion Regulation Scale. It includes for dimensions, namely: Non acceptance, Modulate, Awareness, and Clarity, whose scores range from 1 to 5, where higher scores indicate higher difficulties in the corresponding dimension.

OTHER OUTCOMES:
Interoceptive accuracy before the negative mood induction procedure | The whole study is conducted in a single experimental session: Immediately before the negative mood induction procedure
  Heartbeat Counting Task. Scores range from 0 to 1, with higher scores indicating higher interoceptive accuracy.
Interoceptive sensibility before the negative mood induction procedure | The whole study is conducted in a single experimental session: Immediately before the negative mood induction procedure
  Multidimensional Assessment of Interoceptive Awareness-2. It assesses the following eight dimensions: Noticing, Not-Distracting, Not-Worrying, Attention Regulation, Emotional Awareness, Body Listening, and Trusting. Scores on these dimensions range from 0 to 5, where higher scores indicates higher levels of the corresponding dimension.
Trait difficulties in emotion regulation | The whole study is conducted in a single experimental session: Immediately before the negative mood induction procedure
  Difficulties in Emotion Regulation Scale. It assesses five dimensions, namely: Lack of Emotional Awareness, Nonacceptance of Emotional Responses, Lack of Emotional Clarity, Difficulties Engaging in Goal-Directed Behavior, and Lack of Emotional Control. Scores range from 1 to 5, with higher scores indicating higher difficulties in the corresponding dimension of ER.

CONTACTS AND LOCATIONS:
Overall Officials: Rosa M Baños, PhD, Principal Investigator — Univeristy of Valencia
Locations (3):
- Spain (3):
  - Neurorrehabilitation Service of Hospital VIthas Aguas Vivas, Carcaixent, Valencia
  - Neurorrehabiltiation Service of Hospital Vithas Virgen del Consuelo, Valencia, Valencia
  - Faculty of Psychology and Speech Therapy, University of Valencia, Valencia, Valencia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Baños, R. M., Liaño, V., Botella, C., Alcañiz, M., Guerrero, B., & Rey, B. (2006). Changing Induced Moods Via Virtual Reality. In W. Ijsselsteijn, Y. de Kort, C. Midden, B. Eggen, & E. van den Hoven (Eds.), Persuasive technology. Lecture notes in computer science (pp. 7-15). Springer-Verlag. https://doi.org/10.1007/11755494_3
- [Background] Velten E Jr. A laboratory task for induction of mood states. Behav Res Ther. 1968 Nov;6(4):473-82. doi: 10.1016/0005-7967(68)90028-4. No abstract available. PMID 5714990
- [Background] Lang, P. J., Bradley, M. M., & Cuthbert, B. N. (1999). International affective picture system (IAPS). Instruction manual and affective ratings. The Center for Research in Psychophysiology, University of Florida
- [Background] Eich, E., & Metcalfe, J. (1989). Mood dependent memory for internal versus external events. Journal of Experimental Psychology: Learning, Memory, and Cognition, 15(3), 443-455. https://doi.org/10.1037/0278-7393.15.3.443
- [Background] Sanz, J. (2001). An instrument to evaluate the efficacy of mood induction procedures: The Scale for Mood Assessment. Análisis y Modificación de Conducta, 27(111), 71-110.
- [Background] Lavender JM, Tull MT, DiLillo D, Messman-Moore T, Gratz KL. Development and Validation of a State-Based Measure of Emotion Dysregulation. Assessment. 2017 Mar;24(2):197-209. doi: 10.1177/1073191115601218. Epub 2016 Jul 27. PMID 26297011
- [Background] Katz BA, Lustig N, Assis Y, Yovel I. Measuring regulation in the here and now: The development and validation of the State Emotion Regulation Inventory (SERI). Psychol Assess. 2017 Oct;29(10):1235-1248. doi: 10.1037/pas0000420. Epub 2016 Dec 12. PMID 27936820
- [Background] Pollatos O, Herbert BM, Mai S, Kammer T. Changes in interoceptive processes following brain stimulation. Philos Trans R Soc Lond B Biol Sci. 2016 Nov 19;371(1708):20160016. doi: 10.1098/rstb.2016.0016. Epub 2016 Oct 10. PMID 28080973
- [Background] Mehling WE, Acree M, Stewart A, Silas J, Jones A. The Multidimensional Assessment of Interoceptive Awareness, Version 2 (MAIA-2). PLoS One. 2018 Dec 4;13(12):e0208034. doi: 10.1371/journal.pone.0208034. eCollection 2018. PMID 30513087
- [Background] Gratz, K. L., & Roemer, L. (2004). Multidimensional assessment of emotion regulation and dysregulation: Development, factor structure, and initial validation of the difficulties in emotion regulation scale. Journal of Psychopathology and Behavioral Assessment, 26(1), 41-54.
- [Background] Hervás, G., & Jódar, R. (2008). The Spanish version of the difficulties in emotion regulation scale. Clínica y Salud, 19(2), 139-156.
- [Background] Terol-Cantero, M. C., Cabrera-Perona, V., & Martín-Aragón, M. (2015). Hospital Anxiety and Depression Scale (HADS) review in Spanish samples. Anales de Psicología, 31(2), 494-503. https://doi.org/10.6018/analesps.31.2.172701
- [Background] Zigmond AS, Snaith RP. The hospital anxiety and depression scale. Acta Psychiatr Scand. 1983 Jun;67(6):361-70. doi: 10.1111/j.1600-0447.1983.tb09716.x. PMID 6880820